CLINICAL TRIAL: NCT02848235
Title: Implementing the PMTCT Standard of Care Under Routine Conditions With and Without the Enhanced Mentor Mother ProgrAm (EMMA): A Site-randomized Impact Evaluation Study Among Maternal and Child Health Clinics Supported by the South Rift Valley PEPFAR Program in Kenya
Brief Title: Kenya Enhanced Mentor Mother ProgrAm (EMMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Kenya Ministry of Health (Other Government); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RV 465/WRAIR 2330/EMMA Study
Record Dates: First submitted 2016-07-19; First posted 2016-07-28 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: HIV; Pregnancy
Keywords: Prevention of Mother to Child Transmission; Antenatal Care for HIV positive women; Kenya
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Standard of Care) (No Intervention): Participants in group 1 will receive the standard of care for the Prevention of Mother to Child Transmission (PMCTC) of HIV from the clinic's Mentor Mothers.
- Group 2 (Standard of Care + EMMA) (Experimental): Participants in group 2 will receive the standard of care for Prevention of Mother to Child Transmission (PMCTC) of HIV plus study-specific enhanced care interventions from the clinic's Mentor Mothers.
  Interventions: Other: Standard of Care + EMMA

INTERVENTIONS:
Other: Standard of Care + EMMA — Mother Mentors will provide enhanced care, above that of the standard of care, to include clinic visit exit discussions, visit reminder messages, and patient follow-up in the event that a clinic visit is missed.
  Arms: Group 2 (Standard of Care + EMMA)

SUMMARY:
Kenya recently adopted new treatment guidelines for pregnant women with HIV, which calls for all women to initiate triple-drug antiretroviral therapy (ART) at or soon after their first visit for antenatal care. As part of this new standard of care to prevent mother to child transmission of HIV (PMTCT), Kenya also established the Kenya Mentor Mother Program (KMMP) in 2012 to provide guidance for standardizing peer education and psychosocial support services within the national PMTCT program. This new standard of care (life-long ART and the KMMP) will only yield significant improvements in preventing mother to child transmission if women accept the triple-drug treatment during pregnancy and adhere to visit schedules so that they receive uninterrupted supplies of their medications during pregnancy through at least the cessation of breastfeeding. The primary objectives of this study are: (1) to evaluate implementation of the new guidelines in Kenya under actual, real-world conditions in major maternal and child health clinics in the southern Rift Valley region of Kenya; and (2) to evaluate, also under routine program conditions, the benefits of an innovative intervention package designed to improve implementation of the new treatment guidelines. The intervention uses the existing Mentor Mothers, who already are part of the PMTCT program staff at clinics. At the end of each clinic visit, the Mentor Mother will review with patients their treatment plan and schedule their next visit. The Mentor Mother will also offer, at each encounter, to send a text message reminder to the patient for their next clinic visit and offer to set up an automatic reminder directly on the patient's cell phone. The intervention strategy was developed in close collaboration with local health facility and PMTCT program staff based on their prior and on-going experience providing PMTCT services in the region, and this strategy has the potential to dramatically improve PMTCT service delivery and support global goals to eliminate mother to child transmission.

The study is taking place in 12 clinics in the south-rift valley region of Kenya. A total of 360 patients will be enrolled into the study (approximately 30 at each clinic). The investigators are enrolling patients to receive their permission to look at information recorded in their medical records. All patients eligible for the study, who provide written consent, will be included in the study until the target number of 360 is obtained. After consenting, the study will have no further contact with patients. Because the study only reviews information in medical files that clinics already collect as part of routine care, risks to patients are minimal. The only possible risk is the accidental disclosure of HIV status, but the study is designed to minimize such a risk. There are no direct benefits to study participants, as the study is designed to understand existing adherence to PMTCT care and treatment and to improve such adherence. The study is expected to start in 2016 and end in 2019.

DETAILED DESCRIPTION:
Treatment guidelines for women with HIV during pregnancy and after delivery in resource-constrained settings changed significantly with the WHO 2013 guidelines, which recommended that all pregnant women with HIV should initiate triple-combination ART (Option B). With these guidelines, women previously eligible for life-long ART at initiation should continue for life, while the rest should remain on ART at least through the duration of breastfeeding. A related recommendation was that all pregnant women newly diagnosed with HIV should initiate ART as lifelong treatment. As of 2014, the Kenyan Ministry of Health (MOH) recommends Option B+, which includes the "immediate initiation of life-long ART in pregnant and breastfeeding women upon HIV diagnosis with continuous adherence support" regardless of CD4 count. Throughout this document, the 2014 policy is referred to as standard of care (SOC).

Recognizing the barriers pregnant women newly diagnosed with HIV during antenatal care would face if they were referred elsewhere for HIV care and treatment, in 2005 the South Rift Valley PEPFAR program established a policy to integrate all HIV-related care including ART into PMTCT services provided at the larger MCH clinics within the region. As of 2013, this policy began to be implemented in the 12 largest facilities in the program accounting for more than 85% of women newly diagnosed with HIV during pregnancy in the region.

As part of the standard of care, Kenya also developed the National Guidelines for PMTCT Peer Education and Psychosocial Support in Kenya: The Kenya Mentor Mother Program (KMMP). Mentor Mothers are clinic staff members who are also women living with HIV. They are trained and employed to be part of the clinic's medical team to provide pre-test group education sessions, one-on-one and couples counseling, support groups and defaulter tracing. As part of their routine clinic activities, Mentor Mothers obtain consent from their clients for various forms to follow up, including full consent for both phone and SMS follow up (or only phone follow up, or no follow up) as well as consent for home follow up by her or a community health worker.

Successful implementation of the PMTCT services requires that: (1) pregnant women with HIV initiate life-long ART with minimal delay after their first ANC visit (and women already on ART should continue on ART); (2) they continue on treatment through delivery; (3) they continue on treatment after delivery and the cessation of breastfeeding (and continuing for life for their health); and (4) their child completes HIV testing at 6, 36, and 72 weeks so that they are known to be uninfected after the cessation of breast feeding. Kenya does not yet know if the new policy will lead to better PMTCT outcomes, much less how much better, than under the old policy. Information continues to be lacking in Kenya and elsewhere on the ability of PMTCT programs to initiate pregnant women with HIV on ART during pregnancy and retain them on treatment along the PMTCT cascade of care through delivery, cessation of breastfeeding and for the longer term. This information is largely lacking for the time period when countries implemented prior PMTCT policies (e.g., Option A), and such information does not yet exist for the new policy in Kenya.

What information exists suggests significant room for improvement. For example, a recently published study from a treatment program in western Kenya, with an active outreach department, reported that 32% of women initiated on ART during pregnancy disengaged from treatment before delivery. Although the data for this study were from 2006-2009, they indicate the difficulties with retaining pregnant women on ART during pregnancy. Information on other key outcomes, such as the proportion of those eligible who actually initiated treatment are not reported. Another study from roughly the same region of Kenya during the same time period reported that 38% of women newly diagnosed with HIV during pregnancy did not register in the PMTCT program. In two hospitals between Kericho and Nairobi (Gigil and Naivasha), only 4% of women eligible for ART initiated treatment within six months of their HIV diagnosis.

Some evidence suggests that integration of ART within MCH clinics improves linkage to and initiation of treatment. For example, a study from Zambia found that integration of PMTCT including ART into MCH services increased the percentage of women who initiated PMTCT care (44% compared to 25%) and increased the percentage of those eligible who initiated treatment during pregnancy (32% compared to 4%). While integration improved upon these basic outcomes, more than the majority of patients still did not initiate PMTCT care or initiate ART if eligible. Early evidence on the implementation of life-long ART for pregnant women from Malawi suggests that eliminating CD4 counts as an eligibility criterion might facilitate initiation, but some significant share may still not agree to initiate ART, and retention on treatment during and after delivery may remain problematic without specific attention directed towards these issues.

To support effective implementation of then Kenya PMTCT SOC in the South Rift Valley, other regions of Kenya, and in other resource limited settings, better and up-to-date information remains needed on implementation as currently provided in the study region. And recognizing the importance of both timely initiation and retention on treatment during and after pregnancy, active strategies for retaining patients in care are preferable to after-the-fact follow up to re-engage a patient in care who previously disengaged. Thus, feasible programmatic interventions can support successfully implementation of the SOC and long-term patient care beyond pregnancy.

The study proposed here is designed to fill this information gap and to improve implementation of the Kenyan PMTCT SOC. The investigators will evaluate the impacts and costs of an innovative strategy to improve implementation of the SOC. The strategy, called the Enhanced Mentor Mother ProgrAm (EMMA), provides specific structure to the use of Mentor Mothers within PMTCT programs. The EMMA strategy was developed in collaboration with local health facility and PMTCT program staff based on their experience providing PMTCT services within the integrated ART-MCH facilities. If successful, this approach has the potential to improve dramatically PMTCT service delivery and support global goals to eliminate mother to child transmission. This enhancement to the existing Mentor Mother program is consistent with the KMMP guidelines, which emphasize that "The National Guidelines do not intend to remove the space for creativity and innovation in these approaches. On the contrary, the MOH hopes to inspire ongoing dialogue about quality improvements from the clearly defined starting point outlined herein".

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Pregnant women with HIV presenting for antenatal care at a study site
* The ability to understand and the willingness to sign/mark a written informed consent document in English or Kiswahili during 1st or 2nd visit for antenatal care at a study site.

Exclusion Criteria:

* Indication that patient does not intend to receive further antenatal, postnatal, or PMTCT care at the site.
* Patient is not physically and/or emotionally able to complete the informed consent process to initiate/participate in study (mentally ill, drug abuse, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Patient adherence to anti-retroviral therapy (ART) and retention to care | From date of ART initiation to date of next clinic visit until 72 (+/- 4) weeks post-pardum
  Proportion of pregnant women with HIV receiving an uninterrupted supply (enough medication for each day) of ART from treatment initiation to the next clinic visit, clinic visit to clinic visit, etc. until 72 (+/- 4) weeks post-pardum. Potential for adherence to ART and retention to care (assessed by clinic visit attendance) will be evaluated with this information.

SECONDARY OUTCOMES:
Proportion of patients initiating ART within 30 days of their first antenatal care (ANC) visit | 30 days after the first ANC visit
  The proportion of women initiating ART within 30 days of their first ANC visit will be assessed via prescriptions written as noted in medical records.
Proportion of HIV-exposed infants with known HIV results at 72 (+/- 4) weeks post-pardum | 72 (+/- 4) weeks post-pardum
  Kenyan PMTCT guidelines recommend HIV testing for HIV-exposed babies at 6 weeks, 9 months, and 18 months (72 weeks) of life. Thus, all infants should have a final HIV diagnosis by 72 weeks (either negative at 72 weeks or positive at or before 72 weeks). From the perspective of the clinic, it is critical to getting care to all HIV-infected children that all HIV-exposed babies get a final HIV diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Sawe, MBChB, MMED, Principal Investigator — KEMRI/WRP
Locations (12):
- Kenya (12):
  - Bomet Health Centre, Bomet
  - Kapsabet District Hospital, Kapsabet
  - Kapkatet District Hospital, Kericho
  - Kericho District Hospital, Kericho
  - Bodi Health Centre, Kisumu
  - Munyuanda Health Centre, Kisumu
  - Ratta Health Centre, Kisumu
  - Kombewa County Hospital, Kombewa
  - Longisa District Hospital, Longisa
  - Meteitei-Sub-district Hospital, Nandi Hills
  - Nandi Hills District Hospital, Nandi Hills
  - Transmara District Hospital, Narok

REFERENCES:
- [Result] Larson BA, Tsikhutsu I, Bii M, Halim N, Agaba P, Sugut W, Muli J, Sawe F. The effects of revised peer-counselor support on the PMTCT cascade of care: results from a cluster-randomized trial in Kenya (the EMMA study). BMC Infect Dis. 2023 Apr 25;23(1):257. doi: 10.1186/s12879-023-08246-4. PMID 37098468
- [Result] Larson BA, Halim N, Tsikhutsu I, Bii M, Coakley P, Rockers PC. A tool for estimating antiretroviral medication coverage for HIV-infected women during pregnancy (PMTCT-ACT). Glob Health Res Policy. 2019 Oct 15;4:29. doi: 10.1186/s41256-019-0121-3. eCollection 2019. PMID 31637308
- [Derived] Larson BA, Bii M, Tsikhutsu I, Halim N, Wolfman V, Coakley P, Sugut W, Sawe F. The Enhanced Mentor Mother ProgrAm (EMMA) for the prevention of mother-to-child transmission of HIV in Kenya: study protocol for a cluster randomized controlled trial. Trials. 2018 Oct 30;19(1):594. doi: 10.1186/s13063-018-2975-y. PMID 30376872